CLINICAL TRIAL: NCT01589653
Title: A 20-week Study Comparing Patient-adjusted Versus Physician-adjusted Titration of BIAsp 30 Combined With Metformin in Type 2 Diabetes Patients Uncontrolled on NPH Insulin
Brief Title: Comparing Patient-adjusted Versus Physician-adjusted Titration of BIAsp 30 Combined With Metformin in Type 2 Diabetes Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-3968; U1111-1125-7572 (Other: WHO)
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Results first posted 2016-08-09 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subject-driven titration (Experimental)
  Interventions: Drug: biphasic insulin aspart 30
- Investigator-driven titration (Experimental)
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Dose individually adjusted by the subjects themselves according to the titration algorithm every second week. Administered subcutaneously (s.c., under the skin) twice daily.
  Arms: Subject-driven titration
Drug: biphasic insulin aspart 30 — Dose individually adjusted according to the directions given by the investigator. Administered subcutaneously (s.c., under the skin) twice daily.
  Arms: Investigator-driven titration

SUMMARY:
This trial is conducted in Africa and Asia. The aim of the trial is to compare patient-adjusted versus physician-adjusted titration of BIAsp 30 combined with metformin in type 2 diabetes patients uncontrolled on NPH insulin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for a minimum of 12 months prior to screening
* Currently treated with a NPH insulin for at least 3 months prior to screening
* Stable treatment (no change in dose or regimen) with a total daily dose of at least 1500 mg metformin or maximum tolerated dose (minimum 1000 mg) ± additional OAD treatment. The metformin treatment must have been stable for at least 2 months prior to screening
* HbA1c between 7.0% and 10.0% (both inclusive). (One re-test within one week of screening visit is allowed. The last sample will be conclusive.)
* Body Mass Index (BMI) below or equal to 40.0 kg/m^2
* Able and willing to eat at least 2 main meals each day during the trial
* Able and willing to adhere to the protocol including compliance with performance of self measured plasma glucose (SMPG), injection regimen and titrating themselves according to the protocol
* Experience in performing self-measured plasma glucose (SMPG)

Exclusion Criteria:

* Treatment with any thiazolidinedione (TZD) and Glucagon-like peptide-1 (GLP-1) receptor agonists or pramlintide within the last 3 months prior to screening
* Impaired hepatic function defined as alanine aminotransferase (ALAT) above or equal to 2.5 times upper referenced limit. (One re-test within one week of screening visit is allowed. The last sample will be conclusive.)
* Impaired kidney function with serum creatinine above or equal to 133 µmol/L (1.5 mg/dL) for males and above or equal to 124 µmol/L (1.4 mg/dL) for females. (One re-test within one week of screening visit is allowed. The last sample will be conclusive.)
* Cardiac problems or uncontrolled treated/untreated severe hypertension (defined as systolic blood pressure above or equal to 180 mmHg and/or diastolic blood pressure above or equal to 100 mmHg)
* Previous use of pre-mixed insulin products (pre-mixed insulin analogues or pre-mixed human preparations)
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic episode, during the last 12 months) or hypoglycaemic unawareness as judged by the Investigator or hospitalisation for diabetic ketoacidosis during the previous 6 months
* Known proliferative retinopathy or maculopathy requiring treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2012-05-26 (Actual); Primary Completion 2015-07-09 (Actual); Study Completion 2015-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (13):
- Egypt (3):
  - Novo Nordisk Investigational Site, Alexandria
  - Novo Nordisk Investigational Site, Banī Suwayf
  - Novo Nordisk Investigational Site, Cairo
- Indonesia (2):
  - Novo Nordisk Investigational Site, Bandung
  - Novo Nordisk Investigational Site, Malang
- Morocco (2):
  - Novo Nordisk Investigational Site, Casablanca
  - Novo Nordisk Investigational Site, Marrakesh
- Saudi Arabia (3):
  - Novo Nordisk Investigational Site, Jeddah
  - Novo Nordisk Investigational Site, Riyadh
  - Novo Nordisk Investigational Site, Ta'if
- Novo Nordisk Investigational Site, Tunis, Tunisia
- Vietnam (2):
  - Novo Nordisk Investigational Site, Hà Nội
  - Novo Nordisk Investigational Site, Ho Chi Minh City

REFERENCES:
- [Result] Chraibi A, Al-Herz S, Nguyen BD, Soeatmadji DW, Shinde A, Lakshmivenkataraman B, Assaad-Khalil SH. An RCT Investigating Patient-Driven Versus Physician-Driven Titration of BIAsp 30 in Patients with Type 2 Diabetes Uncontrolled Using NPH Insulin. Diabetes Ther. 2017 Aug;8(4):767-780. doi: 10.1007/s13300-017-0268-1. Epub 2017 May 18. PMID 28523482
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 18 sites in 5 countries as follows: Egypt: 4 sites, Indonesia: 2 sites, Morocco: 4 sites, Saudi Arabia: 4 sites, Vietnam: 4 sites.
Pre-assignment Details: The subjects continued on their previous NPH insulin and OADs upto randomisation (visit 2). At randomisation, the subjects discontinued these treatments except metformin.
Groups:
- Subject-driven Titration: The subjects received BIAsp 30. The treatment dose was individually adjusted by the subjects themselves according to the titration algorithm every second week. Trial product was administered subcutaneously (s.c., under the skin) twice daily.
- Investigator-driven Titration: The subjects received BIAsp 30. The treatment dose was adjusted according to the directions given by the investigator. Trial product was administered subcutaneously (s.c., under the skin) twice daily.
Period: Overall Study
Arm/Group | Subject-driven Titration | Investigator-driven Titration
Started | 76 | 79
Exposed | 76 | 78
Completed | 69 | 68
Not Completed | 7 | 11
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal criteria | 4 | 7
Not completed — Unclassified | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subject-driven Titration | Investigator-driven Titration | Total
Number analyzed (Participants) | 76 | 79 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (10.22) | 54.9 (9.77) | 54.7 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 56 | 116
  Male | 16 | 23 | 39
HbA1c (%) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.5 (0.88) | 8.7 (0.78) | 8.6 (0.83)
Fasting plasma glucose (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 156.8 (59.03) | 148.5 (54.24) | 152.6 (56.64)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline
Description: Change in HbA1c (%) from baseline to the end of the treatment period.
Time Frame: Week 0, week 20
Population: Full analysis set (FAS) included all randomised subjects.
Measure: Least Squares Mean (Standard Error); unit: percentage change in HbA1c
Arm/Group | Subject-driven Titration | Investigator-driven Titration
Number analyzed (Participants) | 76 | 79
percentage change in HbA1c | -1.27 (0.11) | -1.04 (0.11)
Statistical Analysis 1: Comparison: Subject-driven Titration vs Investigator-driven Titration; The null-hypothesis was tested against the alternative hypothesis of non-inferiority as given by: H0: D > 0.4% against HA: D ≤ 0.4% where D is the mean treatment difference for change in HbA1c (subject-driven titration minus investigator-driven titration); Test type: Non-Inferiority or Equivalence — Non-inferiority was to be considered confirmed if the upper bound of the two-sided 95% CI was below or equal to 0.4% or equivalently when the p-value for the one-sided test of H0: D > 0.4% against HA: D ≤ 0.4%, was less than or equal to 2.5%, where D is the mean treatment difference (subject-driven titration minus investigator-driven titration); p < 0.001, Regression, Linear; Analyses were adjusted for treatment, strata, country and baseline HbA1c; Treatment difference = -0.23, 95% CI 2-sided [-0.54 to 0.08]

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) (Laboratory Values) From Baseline
Description: Change in FPG (laboratory values) from baseline to the end of the treatment period
Time Frame: Week 0, week 20
Population: Full analysis set (FAS) included all randomised subjects. Missing data were imputed using last observation carried forward (LOCF). A total of 150 subjects contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Subject-driven Titration | Investigator-driven Titration
Number analyzed (Participants) | 75 | 75
mg/dL | -20.0 (67.23) | -9.1 (62.99)

3. Secondary Outcome: Number of Hypoglycaemic Episodes During the Trial From Baseline
Description: The number of hypoglycaemic episodes (a blood glucose level of approximately 2.8 mmol/L [50 mg/dL] or plasma glucose level 3.1 mmol/L [56 mg/dL]) during the trial.
Time Frame: Week 20
Population: Full analysis set (FAS) included all randomised subjects. Missing data were imputed using last observation carried forward (LOCF). 154 subjects contributed to the analysis.
Measure: Number; unit: episodes
Arm/Group | Subject-driven Titration | Investigator-driven Titration
Number analyzed (Participants) | 76 | 78
episodes | 167 | 222

4. Secondary Outcome: Change in Patient Reported Outcomes: Treatment-Related Impact Measures for Diabetes (TRIM-D)
Description: Mean change from baseline in Treatment Related Impact Measure - Diabetes (TRIM-D) scores. The score measured treatment satisfaction which included an overall score as well the subscale scores (daily life, diabetes management, compliance and psychological health). The scores were transformed to a 0-100 scale with higher scores indicating a better health state.
Time Frame: Week 0, week 20
Population: Full analysis set (FAS) included all randomised subjects.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Subject-driven Titration | Investigator-driven Titration
Number analyzed (Participants) | 74 | 78
scores on a scale
  Daily life | 1.9 (21.84) | 3.6 (20.04)
  Diabetes management | 12.7 (22.79) | 6.9 (22.77)
  Compliance | 7.2 (27.69) | 8.9 (19.54)
  Psychological health | 8.4 (23.97) | 6.1 (21.82)
  Total score | 8.2 (16.52) | 6.6 (15.14)

5. Secondary Outcome: Change in Patient Reported Outcomes: Treatment-Related Impact Measures for Diabetes (TRIM-D)-Treatment Burden
Description: Mean change from baseline in Treatment Related Impact Measure - Diabetes (TRIM-D) scores. The score measured treatment satisfaction which included a subscale score -treatment burden. The scores were transformed to a 0-100 scale with higher scores indicating a better health state.
Time Frame: Week 0, week 20
Population: Full analysis set (FAS) included all randomised subjects.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Subject-driven Titration | Investigator-driven Titration
Number analyzed (Participants) | 73 | 78
scores on a scale | 10.4 (21.00) | 8.0 (22.90)

ADVERSE EVENTS:
Time Frame: Adverse events from the first trial related activity after the subject has signed the informed consent and until post treatment follow-up period.
Description: Safety analysis set - included all subjects receiving at least one dose of BIAsp 30. Subjects in the safety set will contribute to the evaluation "as treated". Safety analysis set included 154 subjects.
Arm/Group | Subject-driven Titration | Investigator-driven Titration
Serious Adverse Events (participants affected / at risk) | 0/76 | 5/78
Other Adverse Events (participants affected / at risk) | 19/76 | 23/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subject-driven Titration (N=76) | Investigator-driven Titration (N=78)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subject-driven Titration (N=76) | Investigator-driven Titration (N=78)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (6) | 5 (7)
Influenza (Infections and infestations) | 6 (6) | 4 (4)
Headache (Nervous system disorders) | 8 (10) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Individual reports by the investigator should not precede the primary manuscript and should always reference the primary manuscript of the trial. Novo Nordisk reserves the right to prior review of such publications and to ask for deferment of publication of individual site results until after the primary manuscript is accepted for publication.